CLINICAL TRIAL: NCT01579318
Title: A Multicenter Phase II Trial of Intratumoral IL12 Plasmid Electroporation in Cutaneous Lymphoma
Brief Title: Phase II Intratumoral IL12 Plasmid Electroporation in Cutaneous Lymphoma
Acronym: CTCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to company resource constraints
Sponsor: OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I120
Record Dates: First submitted 2012-04-15; First posted 2012-04-17 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Cutaneous T Cell Lymphomas (CTCL); Mycosis Fungoides (MF)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Participants received up to 4 cycles of treatment (3 daily treatments on Days 1, 5 and 8, in a 12-week cycle) of intratumoral injection(s) of tavo at a concentration of 1.0 mg/mL (maximum volume of 1 mL/day distributed over 2-4 lesions), followed immediately by electrical discharge around the tumor site resulting in electroporation of plasmid deoxyribonucleic acid (DNA) into tumor cells.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)

INTERVENTIONS:
Biological: Tavokinogene Telseplasmid (tavo) — Patients received intratumoral injection(s) of tavo.
  Other Names: interleukin-12 gene; IL-12 gene; pIL-12; plasmid DNA encoding human interleukin-12; plasmid IL-12
Device: OncoSec Medical System (OMS) — Electroporation via OMS was performed immediately following intratumoral injection of tavo. A sterile applicator containing 6 stainless steel electrodes arranged in a circle were placed around the tumor. The applicator was connected to the OMS power supply and six pulseswere administered to each tumor lesion at the approximate point of tavo injection.
  Other Names: MedPulser

SUMMARY:
A single arm, open label, multi-center, phase 2 study to assess the safety and anti-tumor activity of ImmunoPulse IL-12® in participants with stage IB to IIIB mycosis fungoides. ImmunPulseIL12® is the combination of intrtumoral interleukin-12 gene (also known as tavokinogene telseplasmid [tavo]) and in vivo electroporation-mediated plasmid deoxyribonucleic acid [DNA] vaccine therapy (tavo-EP) administered using the OncoSec Medical System (OMS).

All participants may receive up to four cycles of treatment consisting of three treatment days, Days 1, 5 and 8, in a 12-week cycle as per Protocol version 6 (see Limitations and Caveats section of this record for protocol version information). Patients will receive intra-tumoral injection of tavo at a concentration of 1.0 mg/mL (maximum volume of 1 mL/day distributed over 2-4 lesions), followed immediately by electrical discharge around the tumor site resulting in electroporation of plasmid deoxyribonucleic acid (DNA) into tumor cells.

DETAILED DESCRIPTION:
This is a single arm, open label, multi-center phase 2 study to assess the safety and anti-tumor activity of intratumoral tavo electroporation in participants with stage IB to IIIB mycosis fungoides. All participants received up to four cycles of treatment consisting of three treatment days, Days 1, 5 and 8, in a 12-week cycle. Patients will receive intra-tumoral injection of tavo at a concentration of 1.0 mg/mL (maximum volume of 1 mL/day distributed over 2-4 lesions), followed immediately by electrical discharge around the tumor site resulting in electroporation of plasmid deoxyribonucleic acid (DNA) into tumor cells. Prior to the first cycle of treatment, the investigator will select at least one lesion, or affected area in erythrodermic patients, to be left untreated for the duration of the study to allow for clinical observation of an untreated site. Participants will be followed for safety and clinical evaluation every 4 weeks. Quality of Life will be assessed using the Skindex29, Functional Assessment of Cancer Therapy - General (FACT-G) and Visual Analog Scale for Pruritus (VAS-P) instruments. Survival follow up will occur at 3-month intervals over 2 years following end of study.

ELIGIBILITY:
Inclusion Criteria

1. Biopsy confirmed mycosis fungoides of stage IB - IIIB;
2. Participants must have failed or have been intolerant to at least one standard of care therapy;
3. Participants must have a minimum of one lesion, or affected area in erythrodermic patients (T4/stage III), that meets all following criteria:

   * Accessible for pIL-12 electroporation;
   * Adequate size such that 6-mm biopsy can be collected prior to treatment;
4. Participants must have one additional lesion, or affected area in erythrodermic patients, that remains untreated for the duration of the study;
5. Age ≥ 18 years old;
6. Participants must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
7. Required wash out period of 4 weeks from last dose for the following prior therapies:

   * Topical therapy;
   * Radiotherapy (including photo therapy);
   * Multi-agent chemotherapy;
   * Systemic biological therapy;
   * Histone deacetylase inhibitors (HDAC) inhibitors;
   * Interferon alpha and other investigational therapies;
8. For women of childbearing potential, negative pregnancy serum test within 14 days to the first study drug administration, and use of birth control from 30 days prior to the first day study drug administration and 30 days following last day study drug administration;
9. Male participants must be surgically sterile, or must agree to use contraception during the study and at least 30 days following the last day of study drug administration.
10. Life expectancy of at least 6 months;
11. The patient must have adequate renal and hepatic function as assessed by standard laboratory criteria within 4 weeks prior to enrollment:

    * Creatinine < 2 x upper limit of normal (ULN);
    * Serum bilirubin within institutional normal limits;
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x ULN;
    * Absolute neutrophil count (ANC) > 1000/mm;
    * Platelet count > 100,000 /mm;
12. Able to give informed consent and able to follow guidelines given in the study.

Exclusion Criteria

1. Prior therapy with IL-12 or prior gene therapy;
2. Prior treatment with Campath (alemtuzumab) within 1 year of enrollment;
3. Concurrent immunotherapy, chemotherapy, or radiation therapy for duration of patient participation on study;
4. Concurrent steroid therapy;
5. Concurrent anticoagulant therapy (acetylsalicylic acid [ASA]≤ 325mg/day allowed);
6. Evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study enrollment;
7. Patients with current evidence of large cell transformation (LCT) with aggressive disease at study entry (patients with a history of LCT are eligible if pathologic evidence at study entry indicates there is no presence of LCT);
8. Known history of human immunodeficiency virus (HIV), Human T-cell leukemia virus (HTLV) -1/2 infection, hepatitis B or hepatitis C (active, prior treatment, or both);
9. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 2 years;
10. Significant cardiovascular disease (i.e. New York Heart Association [NYHA] class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias);
11. Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with patient's participation in the study, or to interfere with the interpretation of the results;
12. Participants with electronic pacemakers or defibrillators are excluded from this study as the effect of electroporation on these devices is unknown;
13. Pregnant and breast-feeding women are excluded from the study as effects on the fetus are unknown and there may be a risk of increased fetal wastage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-06-08 (Actual); Primary Completion 2014-06-03 (Actual); Study Completion 2014-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Helen Diller Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 investigative sites in the United States from 08 June 2012 to 03 June 2014.
Period: Overall Study
Arm/Group | Treatment
Started | 2
Completed | 1
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Treatment
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Assessed by Modified Severity Weighted Assessment Tool (mSWAT) Score in the Skin
Description: ORR is defined as the percentage of participants that achieved a complete response (CR) or partial response (PR) as assessed by mSWAT score. The mSWAT defines 3 lesion types and assigns each a weighing factor: patch (no induration or significant elevation)=1; plaque (induration, crusting, ulceration or poikiloderma)=2; tumor (solid or nodular ≥ 1 cm in diameter with evidence of deep infiltration and/or vertical growth)=4. Lesions are assessed by body surface area (BSA) where palm + fingers = approximately 1% BSA in each of 12 areas (head, neck, anterior trunk, arms, forearms, hands, posterior trunk, buttocks, thighs, legs, feet, groin), and the sum of each area of BSA is multiplied by its weighing factor. An overall sum of each subtotal represents the mSWAT score (0=no lesions; 400=lesions covering all areas). CR=100% clearance of skin lesions; PR= 50%-99% clearance of skin disease from baseline without new tumors ( ≥1.0 cm in diameter) in patients with T1, T2 or T4 only skin disease.
Time Frame: Every 28 days for the first 24-weeks of treatment
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 2
percentage of participants | 50.0

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, medical treatment or procedure and which did not necessarily have to have had a causal relationship with this treatment. An adverse event could have, therefore, been any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, medical treatment or procedure whether or not considered related to the medicinal product. An SAE was defined an any untoward medical occurrence that at any dosage resulted in one or more of the following: death, A life-threatening adverse event (real risk of dying), inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly, required intervention to prevent permanent impairment of damage.
Time Frame: From the start of study treatment up to 340 days
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 2
percentage of participants
  AEs | 100.0
  SAEs | 0

3. Secondary Outcome: Duration of Overall Objective Response Assessed by mSWAT Skin Score
Description: Duration of overall objective response (CR or PR) is defined as the number of days from the initial documentation of an objective response to the most current evaluation of that response or to documentation of progression assessed by mSWAT Skin Score: CR=100% clearance of skin lesions; PR= 50%-99% clearance of skin disease from baseline without new tumors ( ≥1.0 cm in diameter) in patients with T1, T2 or T4 only skin disease.
Time Frame: From first documented response until disease progression (Up to 340 days)
Population: All enrolled participants who achieved an objective response.
Measure: Number; unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 1
days | 229

4. Secondary Outcome: Time to Overall Objective Response Assessed by mSWAT Skin Score
Description: Time to overall objective response (CR or PR) is the number of days from the start of therapy to the first documentation of objective response assessed by mSWAT Skin Score: CR=100% clearance of skin lesions; PR= 50%-99% clearance of skin disease from baseline without new tumors ( ≥1.0 cm in diameter) in patients with T1, T2 or T4 only skin disease.
Time Frame: From start of study treatment until overall objective response (Up to 340 days)
Population: All enrolled participants who achieved an objective response.
Measure: Number; unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 1
days | 90

5. Secondary Outcome: Quality of Life (QoL)
Description: Participants were to complete the following QoL assessments prior to clinical evaluations every 4 weeks: Skindex29, FACT-G (Functional Assessment of Cancer Therapy -General) and VAS-P (Visual Analog for Pruritus) questionnaires.
Time Frame: Every 28 days for up to 340 days
Population: Due to early termination of the study QoL data was not collected and reported.
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Immunologic Effects of IL-12 Plasmid Electroporation in Tissue
Description: This outcome measure was erroneously entered as secondary but is truly an exploratory endpoint.
  Planned analyses were:
  1. Transcriptional analysis of interferon pathway activation, antigen presentation and processing machinery (APM) upregulation, and immune cell infiltration in tissue at baseline and post-treatment.
  2. Changes in the characterization of local tissue effects, proportion and phenotype, of intratumoral leukocyte subsets post-treatment.
  3. Changes in T cell receptor clonal expansion and persistence of initial clones post- treatment.
  4. Changes in FOXP3 methylation and quantification of regulatory T cells post- treatment.
Time Frame: 2 years
Population: Due to early termination of the study immunologic effects of IL-12 plasmid electroporation in tissue data was not collected and reported.
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Immunologic Effects of IL-12 Plasmid Electroporation in Peripheral Blood
Description: This outcome measure was erroneously entered as secondary but is truly an exploratory endpoint.
  Planned analyses were:
  1. Changes in the proportion of circulating regulatory and effector T cells in peripheral blood.
  2. Changes in phenotype of leukocyte subsets and T cell receptor clonal expansion
Time Frame: 2 years
Population: Due to early termination of the study immunologic effects of IL-12 plasmid electroporation in peripheral blood data was not collected and reported.
Arm/Group | Treatment
Number analyzed (Participants) | 0

8. Primary Outcome: Objective Response Rate Assessed by Modified Severity Weighted Assessment Tool (mSWAT) Composite Global Score
Description: ORR is defined as the percentage of participants that achieved a complete response (CR) or partial response (PR) as assessed by mSWAT Composite Global Score. This assessment evaluated skin, lymph node, blood and visceral involvement. The response generated in each category was used to determine the Global ORR: CR=complete disappearance of all clinical evidence of disease or, no involvement of disease at baseline through time of response evaluation (NI); PR=regression of measurable disease as follows: 100% clearance of skin lesions, all other categories do not have CR/NI and no category has progressive disease (PD) -OR- 50%-99% clearance of skin disease from baseline without new tumors ( ≥1.0 cm in diameter) in patients with T1, T2 or T4 only skin disease, and if any other category was involved at baseline, at least one has CR/PR and no category has PD.
Time Frame: Every 28 days for the first 24-weeks of treatment
Population: mSWAT Composite Score was not collected and reported due to early termination of the study.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start of study treatment up to 340 days.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=2)
Chills (General disorders) | 1
Pyrexia (General disorders) | 1
Pain (General disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Temperature intolerance (General disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Xerosis (General disorders) | 1

LIMITATIONS AND CAVEATS:
Study enrollment was prematurely terminated under protocol version 6.0. No patients signed informed consent under version 7.0. Two (2) of the targeted 27 patients were enrolled. Thus, a formal statistical analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less